CLINICAL TRIAL: NCT05870449
Title: The Impact of Climate Environment in Different Latitudes on the Occurrence of PICC Complications and Intervention Measures - Prospective, Multicenter, Randomized Controlled Study
Brief Title: The Impact of Climate Environment in Different Latitudes on the Occurrence of PICC Complications
Acronym: PICC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong Branden Med.Device Co.,Ltd (Industry)
Collaborators: Hainan Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: hainan-01
Record Dates: First submitted 2023-05-06; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Cancer; Thrombus; Phlebitis; Infections
MeSH Terms: conditions — Neoplasms; Thrombosis; Phlebitis; Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- trial group (Experimental)
  Interventions: Device: tunneled PICC
- control group (Active Comparator)
  Interventions: Device: routine PICC

INTERVENTIONS:
Device: tunneled PICC — Tunneled PICC is a type of PICC catheterization technique that involves establishing a subcutaneous tunnel to keep the outlet of the catheter away from the puncture site
  Arms: trial group
Device: routine PICC — Peripherally inserted central venous catheterization is a technique that involves inserting PICC through the peripheral vein and infusing drugs into the central vein through a catheter.
  Arms: control group

SUMMARY:
In this study, eligible subjects were randomly assigned to the experimental or control group through randomization (1:1). Under the guidance of electrocardiographic Doppler ultrasound guided puncture and catheterization (EDUG) technology, the tunnel puncture method was compared with the conventional puncture method. The two groups of patients were observed and evaluated intraoperative and postoperative 7 ± 3 days, 30 ± 7 days, 60 ± 10 days, and 90 ± 10 days 120 ± 10 days (if any) and the occurrence of complications during extubation or unplanned extubation at the end of treatment, comparing cases in the north and south, as well as complications related to different catheterization methods

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years old;
* Patients who follow medical advice and require PICC catheterization;
* Patients who have not participated in other clinical studies;
* Patients who voluntarily participate in this clinical study and can cooperate with clinical follow-up;
* There are no serious cardiovascular diseases, such as atrial fibrillation, pulmonary heart disease, and other P-wave abnormalities before catheterization, as well as severe heart conduction block

Exclusion Criteria:

* Known allergies to catheter materials;
* There is a history of infection, injury, and radiation therapy at the puncture site;
* The puncture site has a history of venous thrombosis or surgery;
* Severe abnormal coagulation function;
* Superior vena cava compression syndrome;
* Surgical side limbs of breast cancer patients undergoing radical mastectomy or axillary lymph node dissection;
* Heart pacemaker and arteriovenous fistula on the same side of the limb;
* Patients or patients' family members refuse to sign the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1666 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
rate of complications | 120 days after operation

SECONDARY OUTCOMES:
time of catheter retention | 7, 30, 60, 90 and 120 days after operation

OTHER OUTCOMES:
rate of unplanned extubation | 7, 30, 60, 90 and 120 days after operation
Success rate of one-time catheterization | 7, 30, 60, 90 and 120 days after operation
Operation time | Immediately after operation
incidence of difficulty in pulling out the tube | 7, 30, 60, 90 and 120 days after operation